CLINICAL TRIAL: NCT02011568
Title: Therapeutic Hypothermia Following Out-of-Hospital Cardiac Arrest - A Randomized Trial Comparing Mild and Moderate Therapeutic Hypothermia (CAPITAL CHILL)
Brief Title: Mild Versus Moderate Therapeutic Hypothermia in Out-of-hospital Cardiac Arrest Patients
Acronym: CAPITALCHILL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013106-01
Record Dates: First submitted 2013-11-08; First posted 2013-12-13 (Estimated); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Arrest
Keywords: Therapeutic Hypothermia; Out of hospital cardiac arrest; Mild hypothermia; Moderate hypothermia
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate hypothermia (Other): Therapeutic hypothermia at 31 degrees celsius
  Interventions: Other: Therapeutic Hypothermia
- Mild Hypothermia (Active Comparator): Therapeutic Hypothermia at 34 degrees Celsius
  Interventions: Other: Therapeutic Hypothermia

INTERVENTIONS:
Other: Therapeutic Hypothermia

SUMMARY:
This trial is currently a single-center, randomized, double-blind investigator initiated prospective clinical trial initiated at the University of Ottawa Heart Institute (UOHI). The plan is to expand the trial shortly as a multi-center project. The patients for this study will be recruited amongst comatose survivors of out-of-hospital cardiac arrest (OHCA). The aim of this study is to determine whether neurologic outcomes at six months are improved with moderate (31 degrees Celsius) versus mild (34 degrees Celsius) therapeutic hypothermia (TH) following return of spontaneous circulation (ROSC) in patients suffering OHCA, with ROSC defined as the resumption of sustained perfusing cardiac activity.

The primary outcome will be the proportion of patients experiencing death or a poor neurologic outcome at six months after out of hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

1. Out of hospital cardiac arrest patient
2. Return of spontaneous circulation
3. Glasgow Coma Score equal or lesser than 8.

Exclusion Criteria:

1. Patients residing in a Nursing Home or patients unable to reside independently,
2. Intracranial bleed responsible for the cardiac arrest,
3. Severe coagulopathy with clinical evidence of major bleeding,
4. Coma that is not attributable to cardiac arrest,
5. Pregnancy,
6. Life expectancy of < one year due to any cause unrelated to the cardiac arrest,
7. Known coagulation disorder (i.e. INR >2.0, platelets <100,000 / mm3),
8. Participation in a study with another investigational device or drug < four weeks,
9. The Endovascular cooling (ZOLL) device is not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2013-08; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel R Le May, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Le May M, Osborne C, Russo J, So D, Chong AY, Dick A, Froeschl M, Glover C, Hibbert B, Marquis JF, De Roock S, Labinaz M, Bernick J, Marshall S, Maze R, Wells G. Effect of Moderate vs Mild Therapeutic Hypothermia on Mortality and Neurologic Outcomes in Comatose Survivors of Out-of-Hospital Cardiac Arrest: The CAPITAL CHILL Randomized Clinical Trial. JAMA. 2021 Oct 19;326(15):1494-1503. doi: 10.1001/jama.2021.15703. PMID 34665203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with out-of-hospital cardiac arrest surviving to hospital admission and referred for post-cardiac arrest care were recruited.
Groups:
- Moderate Hypothermia: Therapeutic hypothermia at 31 degrees celsius
  Therapeutic Hypothermia
- Mild Hypothermia: Therapeutic Hypothermia at 34 degrees Celsius
  Therapeutic Hypothermia
Period: Overall Study
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Started | 193 | 196
Completed | 184 | 183
Not Completed | 9 | 13
Not completed — Withdrawal by Subject | 8 | 10
Not completed — Physician Decision | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Hypothermia | Mild Hypothermia | Total
Number analyzed (Participants) | 184 | 183 | 367
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (14.2) | 61.7 (13.3) | 61.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 37 | 69
  Male | 152 | 146 | 298
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 184 | 183 | 367

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Death or Poor Neurologic Outcome at 6 Months
Description: The primary outcome of the study will be death or poor neurologic outcome at six months. Neurologic outcome will be assessed by a specialist in rehabilitation medicine using the Disability Ratings Scale (DRS. Patients will be judged to have had a poor neurologic outcome if the score on the DRS scale is >5.
Time Frame: Six months
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 184 | 183
Participants | 89 | 83

2. Secondary Outcome: Number of Mortality
Description: All cause mortality will be recorded. Mortality will be adjudicated as cardiac versus non-cardiac.
Time Frame: 30 days and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 184 | 183
Participants | 80 | 75

3. Secondary Outcome: Number of Participants With Stroke
Description: Stroke will be classified as hemorrhagic versus non-hemorrhagic.
Time Frame: 30 days and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 184 | 183
Participants
  30 days | 8 | 3
  6 months | 8 | 3

4. Secondary Outcome: Number of Participants With Bleeding
Description: Bleeding will be assessed using the TIMI definition and will be scored as major or minor.
Time Frame: During index hospitalization, up to 40 days
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 184 | 183
Participants | 43 | 36

5. Secondary Outcome: Length of Stay in the Unit
Time Frame: Admission to unit to discharge from unit
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 184 | 183
days | 10 [7 to 15] | 7 [6 to 12]

6. Secondary Outcome: Length of Stay in the Hospital
Description: The length of stay participant was in hospital (day of admission to day of discharge from facility)
Time Frame: Admission to hospital to discharge from hospital.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 184 | 183
days | 22 [16 to 30] | 20 [13 to 36]

7. Secondary Outcome: Number of Participants With Cardiogenic Shock
Description: The total number of participants who had cardiogenic shock during their admission (day of admission to day of discharge from facility)
Time Frame: During index hospitalization - day of admission to day of discharge from the facility (*up to 30 days post admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 184 | 183
Participants | 71 | 61

8. Secondary Outcome: Number of Participants With Repeat Circulatory Arrest Requiring Cardiopulmonary Resuscitation (CPR)
Time Frame: Six months
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 184 | 183
Participants | 20 | 17

9. Secondary Outcome: Number of Participants With Seizures
Description: Count of participants who had seizures while in hospital (day of admission to day of discharge from the facility)
Time Frame: During index hospitalization (*up to 45 days post admission day while in hospital)
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 184 | 183
Participants | 23 | 13

10. Secondary Outcome: Number of Participants With Renal Failure Requiring Renal Replacement Therapy
Description: Participants who required renal replacement therapy (e.g. CRRT, IHD)
Time Frame: During index hospitalization - day of admission up to 45 days post admission while in hospital
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 184 | 183
Participants | 23 | 13

11. Secondary Outcome: Number of Participants With Ventilator Associated Pneumonia
Description: The number of participants who developed ventilator associated pneumonia
Time Frame: During index hospitalization - from day of admission up to 45 days post admission (while in hospital)
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 184 | 183
Participants | 124 | 116

12. Secondary Outcome: Number of Participants With Stent Thrombosis
Description: Participants who are diagnosed with stent thrombosis
Time Frame: Within 6 months of their admission
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 184 | 183
Participants | 2 | 4

13. Secondary Outcome: Number of Participants Discharged Home
Time Frame: Six months
Population: Survivors discharged to home from hospital.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Hypothermia | Mild Hypothermia
Number analyzed (Participants) | 103 | 107
Participants | 93 | 99

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | Moderate Hypothermia | Mild Hypothermia
All-Cause Mortality (participants affected / at risk) | 80/184 | 75/183
Serious Adverse Events (participants affected / at risk) | 28/184 | 34/183
Other Adverse Events (participants affected / at risk) | 0/184 | 0/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Hypothermia (N=184) | Mild Hypothermia (N=183)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 21 (21) | 20 (20)
Inferior Vena cava thrombosis (Blood and lymphatic system disorders) | 7 (7) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-03-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT02011568/Prot_SAP_000.pdf